CLINICAL TRIAL: NCT06133452
Title: Clinical Outcomes of Patients Undergoing Skin-Reducing Mastectomies: A Long-Term Retrospective Study.
Brief Title: Clinical Outcomes of Patients Undergoing Skin-Reducing Mastectomies
Acronym: SRM
Status: Completed | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: UID 4357
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
Keywords: skin reducing mastectomy; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: skin reducing mastectomy — The goal of mastectomy skin reducing is to create a breast reconstruction that appears natural and aesthetically harmonious by minimizing excess skin. Excess skin can be removed in two main ways: as a conventional ellipse around the nipple-areola complex or, preferably, as part of an inverted "T"-shaped incision, commonly used in reduction mammoplasty. This procedure adheres to oncological principles of skin-conserving mastectomy and also incorporates a lower dermal flap, used to create a dermo-muscular pocket that reinforces the coverage of the prosthetic implant.
  This technique allows complete detachment of the pectoral muscle at the bottom while ensuring full coverage of the prosthetic implant with a dermo-muscular layer. By increasing the implant pocket and providing an additional tissue layer at the bottom of the breast, this technique can reduce the risk of complications and improve aesthetic outcomes.

SUMMARY:
The "mastectomy skin reducing" is a surgical procedure involving the removal of the mammary gland and, simultaneously, reducing the excess skin to enhance the aesthetic appearance in breast reconstruction. This technique is commonly used in patients with an excessive amount of residual skin after breast tissue removal, such as following a mastectomy for breast cancer treatment or prophylactic purposes (in patients at high risk of breast carcinoma due to family history and/or mutations in the Breast Cancers genes ).

The goal of mastectomy skin reducing is to create a breast reconstruction that appears natural and aesthetically harmonious by minimizing excess skin. Excess skin can be removed in two main ways: as a conventional ellipse around the nipple-areola complex or, preferably, as part of an inverted "T"-shaped incision, commonly used in reduction mammoplasty. This procedure adheres to oncological principles of skin-conserving mastectomy and also incorporates a lower dermal flap, used to create a dermo-muscular pocket that reinforces the coverage of the prosthetic implant.

The primary indication for mastectomy skin reducing is when a patient has excessively large (hypertrophic) and sagging (ptotic) breasts. In these cases, removing excess skin and breast tissue during mastectomy contributes to creating a solid foundation for breast reconstruction and improving the aesthetics of the reconstructed breast.

The purpose of this retrospective study is to provide accurate data on the clinical outcomes of mastectomy skin reducing performed at the European Oncology Institute in Milan. This study is part of a larger project involving patients with breast cancer and/or carriers of mutations in the Breast Cancer genes who have undergone mastectomy skin reducing in the last 5 years.

DETAILED DESCRIPTION:
It is a single-center study, conducted exclusively at the European Oncology Institute ( IEO). It is a retrospective study, analyzing events that occurred in the past. The results of this study, aggregating data from numerous patients, could influence public health policies by improving the efficiency and effectiveness of surgical treatments for patients with breast cancer and/or carriers of Breast Cancers mutations.

The study is independent and non-profit, conducted by a group with no financial interests, and will collect, in addition to genetic data, clinical and pathological information (related to the disease), information on the types of treatments performed, the presence or absence of recurrences or other tumors, and the survival status of patients.

IEO patient data will be transferred in anonymized form (the Oxford group cannot identify patients; only IEO can identify them) using a secure transmission channel. The study has been evaluated and authorized by an independent "Data Governance Board for Retrospective Studies at IEO" considering the scientific relevance of the study and its partners, relevance to the Institute's research lines, and the risk-benefit ratio from scientific, ethical-moral, and personal data protection perspectives.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer affected women with moderate-large Breast underwent to skin reducing mastectomy.
* High risk breast cancer ( BRCA1 and/or 2 mutated) women with moderate-large Breast underwent to skin reducing mastectomy.

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: breast cancer affected and/or High risk breast cancer ( BRCA1 and/or 2 mutated) women with moderate-large Brest underwent to skin reducing mastectomy.
Sampling Method: Non-Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2018-01-07 (Actual); Primary Completion 2023-04-02 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
rate of short term complications | 60 months
  hematoma, seroma, bleeding, infections, necrosis, prothesis exposure,Prothesis Explantations
rate of long term complications | 60 months
  Seroma, Infections, Necrosis, Prothesis Explantations,prothesis exposure

SECONDARY OUTCOMES:
rate of refinements | 60 months
  re-intervention needed

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Vittorio Emanuele Lisa, MD, Principal Investigator — Istituto Europeo di Oncologia
Locations (1):
- Istituto Europeo di Oncologia, Milan, Lombardy, Italy